CLINICAL TRIAL: NCT00771108
Title: Exercise Dose and Nonalcoholic Fatty Liver Disease
Acronym: ED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 06-0039; #5P30 DK052574 (NIH/DDRCC); R01 DK37948 (NIH/NIDDK); R01DK037948 (NIH); 5P30DK052574 (NIH)
Record Dates: First submitted 2008-10-09; First posted 2008-10-13 (Estimated); Last update posted 2011-09-07 (Estimated); Status verified 2011-09

CONDITIONS: Non-alcoholic Fatty Liver Disease (NAFLD)
Keywords: NAFLD; Obesity; Metabolic Syndrome; Nonalcoholic Fatty Liver Disease
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Obesity; Metabolic Syndrome | interventions — Exercise; Walking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- control (No Intervention): Subjects will serve as controls, continuing current diet and activity levels. Subjects will get monthly weights by the investigator at the research center.
- Exercise (Experimental): For 16 weeks subjects will exercise from 30-60 minutes five times a week.
  Interventions: Behavioral: exercise

INTERVENTIONS:
Behavioral: exercise — For 16 weeks subjects will exercise from 30-60 minutes five times a week.
  Other Names: walking
  Arms: Exercise

SUMMARY:
The purpose of this research is to provide a better understanding of how exercise (walking) affects non-alcoholic fatty liver disease (NAFLD) in overweight people. NAFLD, which is common in obese people, occurs when the liver has too much fat.

DETAILED DESCRIPTION:
Non-alcoholic fatty liver disease (NAFLD) affects about 33% of adults in the United States. The prevalence of NAFLD is four to five times higher in obese than lean persons and is associated with insulin resistance and the metabolic syndrome. Decreasing calorie intake and increasing physical activity has been recommended as primary therapy for NAFLD, but the independent effect of aerobic exercise is unknown. The current exercise guidelines for disease prevention and weight management range from 150 min/wk, recommended by the Centers for Disease Control and the American College of Sports Medicine, to 300 min/wk, recommended by the Institute of Medicine. However, it is not known whether aerobic exercise alone can improve NAFLD, and which recommended dose of exercise might have the most beneficial effects. The purpose of this proposal is to determine the effect of moderate intensity endurance exercise on: 1) hepatic fat content; 2) hepatic lipoprotein kinetics; and 3) plasma inflammatory markers. We hypothesize that aerobic exercise will decrease hepatic fat content, improve VLDL kinetics, and decrease inflammation in a dose-dependent fashion. The results from this study will help determine exercise guidelines for obese patients with NAFLD, and lay the groundwork for future studies evaluating the effects of exercise on metabolic diseases associated with obesity.

This proposal involves conducting a randomized controlled trial that will randomize obese subjects with NAFLD (> 10% hepatic fat content) to one of two groups: Group 1 (Control, no exercise) and Group 2 (Moderate Intensity Aerobic Exercise- 150 min/wk to 300 min/wk of supervised exercise performed at 45-55% of O2 max).

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 with Nonalcoholic Fatty Liver Disease as determined by MRS

Exclusion Criteria:

* Medical History

  * Diabetes
  * Heart Disease
  * Asthma/Lung disease
  * Injury that prevents exercise
* Social history

  * Drinking
  * More than one drink per day
  * Binge drinking on the weekends (more than 3 or 4 drinks per weekend day)
* Smoking
* It's OK if they were a previous smoker, but they need to have quit more than 6 months ago
* Exercise

  * They must exercise less than one hour per week
  * Medications: must be on stable regimen of ANY medication for at least 3 months
* Beta-Blockers

  * Lipid/cholesterol lowering medications:
  * Oral hypoglycemics (anti-diabetes medications - some like metformin are indicated for pre-diabetes)
* Hormone replacement therapy
* If the woman is pre-menopausal, it is OK if she is on birth control as long as she has been on it over 3 months
* Weight history

  * Weight <300 lbs
  * BMI 30 to 45
  * Weight stable - <10lbs weight loss or gain in the last 3 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2006-05; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
The effect of aerobic exercise on: Intrahepatic fat content | 3 years

SECONDARY OUTCOMES:
VLDL-triglyceride (TG) and VLDL-Apolipoprotein B (apoB) kinetics | 3 years
Insulin action in liver (suppression of glucose production), muscle (stimulation of glucose uptake), and adipose tissue (suppression of lipolysis). | 3 years
Plasma markers of inflammation | 3 years
Potential cellular mechanisms responsible for changes in insulin action and inflammation | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Klein, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- [Derived] Sullivan S, Kirk EP, Mittendorfer B, Patterson BW, Klein S. Randomized trial of exercise effect on intrahepatic triglyceride content and lipid kinetics in nonalcoholic fatty liver disease. Hepatology. 2012 Jun;55(6):1738-45. doi: 10.1002/hep.25548. Epub 2012 Apr 25. PMID 22213436